CLINICAL TRIAL: NCT00117052
Title: SENSOR: Study to InvestigatE Cinacalcet TreatmeNt in Haemodialysis Patients With SecOndary HyperparathyRoidism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040143
Record Dates: First submitted 2005-06-30; First posted 2005-07-04 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Secondary Hyperparathyroidism; End Stage Renal Disease
Keywords: Clinical trial; Amgen; Secondary HyperParaThyroidism (SHPT); Dialysis; End Stage Renal Disease (ESRD); KDOQI; Cinacalcet
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Kidney Failure, Chronic | interventions — Cinacalcet

ARMS (2):
- During dialysis visit (Active Comparator): Cinacalcet is given during the dialysis visit
  Interventions: Drug: cinacalcet
- Post-dialysis meal (Active Comparator): Cinacalcet is administered with a post-dialysis meal
  Interventions: Drug: cinacalcet

INTERVENTIONS:
Drug: cinacalcet — All eligible subjects were assigned to receive once daily oral doses of cinacalcet, but were randomised in a 1:1 ratio to receive the drug either with the first meal after dialysis or during the dialysis visit on dialysis days.

SUMMARY:
The purpose of this study is to demonstrate that the efficacy of cinacalcet when co-administered with the first meal after dialysis is comparable (non-inferior) to the efficacy of cinacalcet when administered during the dialysis study visit.

ELIGIBILITY:
Inclusion Criteria: - CKD patients requiring dialysis (HD, HDF, HF) for at least 1 month before enrolment - An iPTH determination within 14 days before randomisation must be greater than or equal to 300 pg/mL (biPTH greater than or equal to 150 pg/mL) - A serum calcium determination (corrected for calcium) within 14 days before randomisation must be greater than or equal to 8.4 mg/dL [2.1 mmol/L] Exclusion Criteria: - Have an unstable medical condition, defined as having been hospitalised, other than for dialysis vascular access revision, within 30 days before day 1, or otherwise unstable in the judgment of the investigator - Are currently breast-feeding - Are performing peritoneal dialysis - Have had a parathyroidectomy in the 3 months before day 1 - Have a gastrointestinal disorder that may be associated with impaired absorption of orally administered medications or an inability to swallow tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 673 (Actual)
Dates: Start 2004-09; Primary Completion 2005-11 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects with PTH less than or equal to 300pg/mL | 21 week dose optimisation phase

SECONDARY OUTCOMES:
Changes in Calcium (Ca), Phosphor (P), Ca X P, KDOQI guidelines, Rate of Nausea and Vomiting Aes | Dose Optimisation phase 21 weeks
Safety of cinacalcet | 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Schaefer RM, Bover J, Dellanna F, Sanz D, Asensio C, Sanchez Gonzalez MC, Gross P, Zani V, Carter D, Jehle PM. Efficacy of cinacalcet administered with the first meal after dialysis: the SENSOR Study. Clin Nephrol. 2008 Aug;70(2):126-34. doi: 10.5414/cnp70126. PMID 18793528
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_38_AMG_073_20040143.pdf
- See also: FDA-approved Drug Labeling — http://www.sensipar.com/